CLINICAL TRIAL: NCT03767582
Title: A Phase I/II Trial of Combination Immunotherapy With Nivolumab and a CCR2/CCR5 Dual Antagonist (BMS-813160) With or Without GVAX Following Chemotherapy and Radiotherapy for Locally Advanced Pancreatic Ductal Adenocarcinomas (PDACs).
Brief Title: Trial of Neoadjuvant and Adjuvant Nivolumab and BMS-813160 With or Without GVAX for Locally Advanced Pancreatic Ductal Adenocarcinomas.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J18163; IRB00190660 (Other: JHMI IRB)
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Pancreatic Ductal Adenocarcinoma (PDAC); Pancreatic Ductal Adenocarcinoma
Keywords: GVAX; Nivolumab; CCR2/CCR5 dual antagonist; Anti-PD-1; Cancer vaccine; Monoclonal antibody; Checkpoint inhibitor; Myeloid modulating agent; Immunotherapy; Neoadjuvant chemotherapy; Stereotactic body radiation therapy; SBRT; Pancreatic cancer; Pancreatic Ductal Adenocarcinoma; PDAC; Locally advanced pancreatic ductal adenocarcinoma; LAPC
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Nivolumab; BMS-813160

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I - GVAX/Nivolumab/CCR2/CCR5 dual antagonist (Experimental)
  Interventions: Radiation: Stereotactic Body Radiation (SBRT); Drug: Nivolumab; Drug: CCR2/CCR5 dual antagonist; Drug: GVAX
- Phase II - Arm A: Nivolumab/CCR2/CCR5 dual antagonist (Experimental)
  Interventions: Radiation: Stereotactic Body Radiation (SBRT); Drug: Nivolumab; Drug: CCR2/CCR5 dual antagonist
- Phase II - Arm B: Nivolumab/GVAX/CCR2/CCR5 dual antagonist (Experimental)
  Interventions: Radiation: Stereotactic Body Radiation (SBRT); Drug: Nivolumab; Drug: CCR2/CCR5 dual antagonist; Drug: GVAX

INTERVENTIONS:
Radiation: Stereotactic Body Radiation (SBRT) — SBRT (6.6 Gy over 5 days) will be administered between 2 to 4 weeks after chemotherapy. (Prior to surgery)
Drug: Nivolumab — Nivolumab (480 mg) will be administered IV over 30 minutes, on day 1 of cycle 1 (within 1 to 2 weeks after SBRT prior to surgery). Post - surgery Nivolumab will be given on Day 1 of cycles 2-5. Cycles are 4 weeks long.
  Other Names: OPDIVO
Drug: CCR2/CCR5 dual antagonist — CCR2/CCR5 dual antagonist (150 mg capsules) will be administered orally twice a day, on days 1-28 of cycle 1 (within 1 to 2 weeks after SBRT prior to surgery). Post - surgery CCR2/CCR5 dual antagonist will be given daily on cycles 2-5. Cycles are 4 weeks long.
  Other Names: BMS-813160
Drug: GVAX — Vaccine (5x10^8 cells) will be administered on day 2 of cycle 1 (within 1 to 2 weeks after SBRT prior to surgery). Post - surgery GVAX will be given on Day 2 of cycles 2-5. Cycles are 4 weeks long. Six intradermal injections every 4 weeks.
  Other Names: PANC 10.05 pcDNA-1/GM-Neo vaccine; PANC 6.03 pcDNA-1/GM-Neo vaccine
  Arms: Phase I - GVAX/Nivolumab/CCR2/CCR5 dual antagonist; Phase II - Arm B: Nivolumab/GVAX/CCR2/CCR5 dual antagonist

SUMMARY:
The purpose of this study is to evaluate if the combination of nivolumab and a CCR2/CCR5 dual antagonist (BMS-813160) with GVAX is safe in patients with locally advanced pancreatic cancer (LAPC) who have received chemotherapy and radiotherapy, and to see if this combination therapy enhances the infiltration of CD8+CD137+ cells in PDACs .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patients with histologically- or cytologically-proven, surgically unresectable, locally advanced pancreatic adenocarcinoma.
* If the patient does not have a diagnostic biopsy that is adequate for review at our institution, the patient must agree to a research core biopsy to be performed at Johns Hopkins.
* If the patient's available imaging is not adequate for review by our institution, the patient must agree to a repeat imaging to be performed at Johns Hopkins.
* Patients cannot have had any prior therapy for the locally advanced pancreatic adenocarcinoma.
* ECOG performance status 0 or 1
* Life expectancy greater than 3 months.
* Able to swallow pills or capsules.
* Patient must have adequate organ function defined by the study-specified laboratory tests.
* Patients must be eligible to receive FOLFIRINOX-based chemotherapy.
* Patients must be willing to be treated with stereotactic body radiation therapy (SBRT) only at Johns Hopkins Hospital.
* Patients must be willing to undergo a core biopsy of the pancreatic cancer.
* Patients must be willing to undergo a biopsy of the pancreatic cancer if the patient is not deemed a surgical candidate during the pre-surgical evaluation.
* Must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Have had non-FOLFIRINOX-based chemotherapy for the pancreatic cancer.
* Have received any anti-neoplastic biologics, vaccines or hormonal treatment, including investigational drugs, within 28 days of the first dose of study.
* History of past treatment with immunotherapy agents prior to initial enrollment into this study (including, but not limited to: IL-2, interferon, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40, anti-CTLA-4 or anti-CCR2/5 drugs).
* Have had prior organ or tissue allograft or allogeneic bone marrow transplantation, including corneal transplants.
* Is currently participating or has participated in a study of an investigational agent or using an investigational device for the treatment of cancer.
* Current use of immunosuppressive medications within 14 days prior to study medications.
* Have received any vaccine within 14 days prior to study medications.
* Receiving growth factors including, but not limited to, granulocyte-colony stimulating factor (G-CSF), GM-CSF, erythropoietin, within 14 days of the first dose of study medication.
* History of any autoimmune disease. Patients with thyroid disease will be allowed.
* Has a history of (non-infectious) pneumonitis or current pneumonitis.
* Has a pulse oximetry < 92% on room air.
* Requires the use of home oxygen.
* Patients with uncontrolled intercurrent illness including, but not limited to, myocardial infarction or stroke/transient ischemic attack within the past 6 months, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* 12-lead electrocardiogram with QRS ≥ 120 msec, except right bundle branch block ; QTcF (QT corrected for heart rate using Fridericia's method) ≥ 480 msec, except right bundle branch block
* Has an active infection requiring systemic therapy.
* Infection with HIV or hepatitis B or C.
* Any concurrent malignancy other than non-melanoma skin cancer, non-invasive bladder cancer, early stage prostate cancer, or carcinoma in situ of the cervix.
* Current or recent (within 3 months of study treatment administration) gastrointestinal disease that could impact the absorption of study treatment.
* Any gastrointestinal surgery that is likely impact upon the absorption of study treatment.
* Inability to tolerate oral medication.
* Unable to have blood drawn.
* Have had surgery within 28 days of the first dose of study medication.
* Prior use of strong/moderate CYP3A4 inhibitors or inducers within 28 days of the first dose of BMS-813160.
* Prior use of Class I antiarrhythmics within 28 days of first dose of study medication.
* Has ascites requiring medical management.
* Presence of duodenal or gastric invasion by the tumor.
* Hypersensitivity reaction to any monoclonal antibody.
* Known allergy or hypersensitivity to study drugs or any of their components of the study arm that participant is enrolling.
* Woman who are pregnant or breastfeeding.
* Patient is unwilling or unable to follow the study schedule for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants experiencing study drug-related toxicities | 3 years
  Number of participants who experienced study drug-related toxicities as defined by CTCAE v5.0
Percentage of participants treated with immunotherapy who achieve an immune response | 3 years
  Percentage of participants who have >80% increase of infiltration of CD8+CD137+ T cells into the pancreatic ductal adenocarcinoma after treatment with immunotherapy compared to baseline before treatment.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Number of months from the time of Cycle 1, Day 1 of immunotherapy until death from any cause
Metastasis free survival (MFS) | 3 years
  Number of months from the time of Cycle 1, Day 1 of immunotherapy until first documented distant metastases on imaging per RECIST 1.1 or death from any cause, whichever occurs first.
Local progression free survival (LPFS) Time | 3 years
  Number of months from the time of Cycle 1, Day 1 of immunotherapy until first documented local progression or relapse from complete response on imaging (using RECIST 1.1 criteria and irRECIST criteria) or death from any cause, whichever occurs first.
Surgical Resectability Rate | 3 years
  Number of participants who are able to undergo successful tumor resection (as defined by R0 and R1 resection).
Pathological Response Rate | 3 years
  Number of participants who have a pathologic complete response as determined by surgical margins and residual disease.
Change in Quality of life score based on EORTC QLQ-C30/Pan26 | Baseline, 3 years
  Change in quality of life from baseline will be evaluated using the European Organization for Research and Treatment of Cancer core questionnaire, pancreatic cancer module (EORTC QLQ-C30/Pan26). The QLQ-C30 includes 30 questions assessing global health status/quality of life, function, and symptoms. The PAN26 module comprises of an additional 26 questions assessing pain, dietary changes, jaundice, altered bowel habit, emotional problems related to pancreatic cancer, and other symptoms (cachexia, indigestion, flatulence, dry mouth, taste changes). The score for each item ranges from 0-100, with a higher score reflecting a better level of functioning, a better quality of life, or a worse level of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Narang, MD, Principal Investigator — Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided